CLINICAL TRIAL: NCT02369523
Title: Periarticular Infusion With Liposomal Bupivacaine or a Ropivacaine Cocktail Versus Continuous Femoral Nerve Catheters for Multimodal Pain Management Following Primary TKA: A Randomized Controlled Trial
Brief Title: Multimodal Pain Management Following Primary TKA
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Adequate enrollment was not reached for this study.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Pelt, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 74975
Record Dates: First submitted 2015-02-05; First posted 2015-02-24 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Pain
Keywords: Primary Total Knee Arthroplasty
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- liposomal bupivacaine (LB) (Exparel) (Active Comparator): Mixture of 50 milliliters (mL) of 0.25% Bupivacaine with epinephrine, 40 mL of sterile saline and 20 mL of Exparel®.
  Interventions: Drug: Exparel
- Ropivacaine cocktail (PIC) (Active Comparator): 400 milligrams (mg) Ropivacaine, 5 mg morphine, and 0.4 mg epinephrine in 100 cc solution
  Interventions: Drug: Ropivacaine cocktail (PIC)
- continuous femoral nerve blocks (cFNB) (Active Comparator): Continuous Femoral Nerve Block- 0.25% Bupivacaine at a rate of 5 ml/hour for 48 Hours.
  Sciatic nerve block - 0.125% bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Exparel — Mixture of 50 mL of 0.25% Bupivacaine with epinephrine, 40 mL of sterile saline and 20 mL of Exparel®.
  Arms: liposomal bupivacaine (LB) (Exparel)
Drug: Ropivacaine cocktail (PIC) — 400 mg Ropivacaine, 5 mg morphine, and 0.4 mg epinephrine in 100 cc solution
  Arms: Ropivacaine cocktail (PIC)
Drug: Bupivacaine — Continuous Femoral Nerve Block- 0.25% Bupivacaine at a rate of 5 ml/hour for 48 Hours.
  Sciatic nerve block - 0.125% bupivacaine
  Arms: continuous femoral nerve blocks (cFNB)

SUMMARY:
The investigators plan to evaluate the length of time to discharge readiness between the groups (continuous femoral nerve blocks (cFNB) vs. liposomal bupivacaine (LB) vs. periarticular infusion cocktails (PIC) following primary total knee arthroplasty (TKA). In addition, the investigators will compare quadriceps strength recovery over time and exploratory variables between the groups.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 40 Years Old
* Scheduled for Primary Total Knee Arthroplasty

Exclusion Criteria:

* Opiate Tolerant (≥60mg/day oral morphine/equivalent for ≥1 week)
* Neuromuscular deficit affecting the lower limbs

  * Peripheral neuropathy
  * Radiculopathy/Sciatica
* Known allergy or intolerance to Bupivacaine or Ropivacaine
* Hepatic Disease
* Renal Disease/Patients needing Dialysis
* Planned unicompartmental knee replacement
* Less than 90 degree of knee flexion preoperatively.
* Patients who lack the capacity to consent or are unwilling to do so
* At the discretion of the PI, patients who may have difficulty complying with standard of care (SOC) followup may also be excluded

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time to Discharge Readiness | Participants will be followed for the duration of hospital stay, an average of 3 days
  Time to discharge readiness will be defined as the time from surgical stop to the time of the 2nd consecutive assessment where all criteria are fulfilled.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pelt, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States